CLINICAL TRIAL: NCT04690296
Title: Ultrasound Guidance Versus Anatomical Landmarks for Subclavian Vein Catheterization: a Prospective Randomized Study
Brief Title: Ultrasound Guidance Versus Anatomical Landmarks for Subclavian Vein Catheterization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Tunis El Manar (Other)
Responsible Party: Principal Investigator, Mechaal Benali, Professor, University Tunis El Manar
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: UTEM USG SCV
Record Dates: First submitted 2020-12-27; First posted 2020-12-30 (Actual); Last update posted 2020-12-30 (Actual); Status verified 2020-12

CONDITIONS: Central Venous Catheterization
Keywords: ultrasound guidance; central venous catheterization; subclavain vein

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- US group (Experimental): a group underwent real time USG-SCV catheterization
  Interventions: Device: cathetherization approach
- LM group (Experimental): a group in whom anatomical LM method was used
  Interventions: Device: cathetherization approach

INTERVENTIONS:
Device: cathetherization approach — real time ultrasound guidance versus anatomical landmarks subcalvain vein catheterization

SUMMARY:
This was a prospective randomized study. After prior approval by the Ethics Committee, we included all patients aged over 18 years- old who were admitted to the intensive care unit (ICU) and who required a central venous catheterization (CVC) outside the emergency's context. Non-inclusion criteria were thrombosis of the vein or coagulopathy. All catheterizations were done by the same non-experimented practitioner. Patients were randomized into two groups according to the catheterization's technique of subclavain vein: real-time long axis ultrasound guidance (US group) and anatomical landmarks ( LM group). The main outcome was success. The secondary outcomes were: success' rate at first puncture, number of punctures, rate of redirections, number of redirections, access's time, preparation and spotting time and rate of complications (arterial puncture, hematoma, pneumothorax, wrong position of the catheter).

Data analysis was performed using the SPSS® software version 20: The Student's "t" test was used to compare the normally distributed quantitative variables, the Mann-Whitney's test for non-normally distributed quantitative variables and the Chi-square and Fisher tests for qualitative data. A value of p <0.05 was considered as statistically significant.

DETAILED DESCRIPTION:
Methods:

Study population:

It was a prospective randomized study, conducted in the ICU after obtaining approval by the local ethics committee.

We enrolled all patients older than 18 years and requiring a CVC in non emergent conditions after obtaining a written informed consent from the patient or trusted person.

The exclusion criteria were the vein thrombosis and the existence of a coagulopathy.

Patients were randomly divided according to computer generated randomized table into twogroups: a group underwent real time USG-SCV catheterization (US group) and a group in whom anatomical LM method was used (LM group).

Methods:

All procedures were performed by the same novice operator trained in CVC placement, each of whom had performed at least 10 catheterization using both techniques on cadavers before standing the study.

All patients were mechanically ventilated, they underwent ultrasound scanning of the infraclavicular area to detect an eventual venous thrombosis and they put in trendelenburg position with a block under the homolateral shoulder.

Techniques:

The anterosuperior region of the chest was prepared in a sterile way for both approach In the LM group, we chose the Aubaniac technique to cannulate the SCV(10) . The needle was inserted 1 cm inferior and laterally to the junction of the medial one-third and lateral two-thirds of the clavicle, it was passed below the clavicle and above the first rib and it was advanced parallel to the floor, through the subclavian muscle, until it entered the subclavian vein.

The intravascular position of the catheter was approved by venous blood's reflux.

In the US group, we chose the infraclavicular approach with long axis view(11). A portable ultrasound unit (Mindray M7®, Shenzhen, China) equipped with a 12 MHz linear transducer was used. The probe was covered with ultrasonic gel and wrapped in a sterile sheath. The first step was to visualize the SCV and the artery in a short axis view. Then, maneuvers of the transducer were performed to expose the axillary vein and in its continuation till the SCV on the longitudinal axis to achieve an optimum plane of catheterization.The probe was handled by the non-dominant hand. The needle was introduced slowly with the dominant hand so that its tip's trajectory could be detected superficially. It was advanced in real-time toward the lumen of the vein, on the longitudinal axis, while it was directed toward the acoustic shadow of the thoracic rib underneath. This leads to minimize the risk of damaging the pleurae and the lung in case of an vein's transfixion. Hence, the needle entered the lumen of the vessel either at the level of the axillary vein or at the level of its medial continuation by the SCV . After that,venous blood returned in the syringe.

In the both technique, the guidewire and the catheter were advanced according to the Seldinger's technique (12).

Chest X-ray was used to evaluate the position of the catheter's tip and to detect pneumothorax. Hematoma was detected by ultrasonography.

Demographic characteristics, presence of risks factors for difficult venous catheterization and side of cannulation were recorded for all patients.

The primary outcome was the successful insertion of the catheter. Failure was defined by a number of attempts greater than or equal to five.

The secondary and comes were: the success's rate in the first attempt, the number of attempts, redirections rate, number of redirections, access time (defined as the time between the skin puncture and the return of venous blood) and complications such as hematoma, pneumothorax, arterial puncture and malposition.

Statistical analysis:

Sample size was calculated assuming a difference of proposition of success rate at 20% with a statistical power of 0.85 (alpha = 0.05). The precise sample size estimation was 33 per group and 66 in totals.

Statistical analysis were performed using SPSS 200 software. Normal distributions of continuous variables were compared using Student t-test .Mann-Whitney U test was used for continuous variables without normal distribution. Categorical variables were compared using the χ2 test and Fisher exact test. Data were expressed as mean ± SD or as median (25th percentile - 75th percentile). A p value (two-sided in all tests) of 0.05 was considered significant. A linear regression was used to evaluate the relation between access's time and patient's range.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted in intensive care unit requiring a central venous catheter (CVC)

Exclusion Criteria:

* • Major blood coagulation disorders,

  * Any thrombotic formations within the vein,
  * Congenital or acquired deformity of neck or clavicle
  * Cannulation site infection, hematoma and surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2015-01-05 (Actual); Primary Completion 2015-06-20 (Actual); Study Completion 2015-06-20 (Actual)

PRIMARY OUTCOMES:
the successful insertion of the catheter. | During the venous cannulation procedure
  Failure was defined by a number of attempts greater than or equal to five

SECONDARY OUTCOMES:
the success's rate in the first attempt | During the venous cannulation procedure
  the success's rate in the first attempt
The evolution of the blood reflux time (success) as a function of the rank of the patients in the 02 groups | During the venous cannulation procedure
  procedures were performed by the same novice operator trained in CVC placement.we studied the relationship between the rank of patients and the success rate

CONTACTS AND LOCATIONS:
Overall Officials: mechaal benali, PROFESSOR, Principal Investigator — university manar Tunis tunisia